CLINICAL TRIAL: NCT05257122
Title: A Phase II Clinical Trial of the Safety and Efficacy of Fruquintinib in Advanced Pancreatic Cancer Patients Who Failed Second-line Gemcitabine or 5-FU Based Chemotherapy
Brief Title: A Phase II Clinical Trial of Fruquintinib as Third Line Treatment in Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Collaborators: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Weijian Guo, Proferssor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDZL-FPcT
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Advanced Pancreatic Carcinoma
Keywords: advanced pancreatic carcinoma; fruquintinib; target therapy
MeSH Terms: interventions — HMPL-013

STUDY DESIGN:
Intervention Model Description: This study is an open Label, non-randomized, single-arm and multi-centered phase II clinical trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm A (Experimental): Monotherapy of Fruquintinib
  Interventions: Drug: Fruquintinib

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib 5mg qd, d1-21, q28d
  Other Names: F

SUMMARY:
A Phase II Clinical Trial of the Safety and Efficacy of Fruquintinib in Advanced Pancreatic Cancer Patients Who Failed Second-line Gemcitabine or 5-FU Based Chemotherapy

DETAILED DESCRIPTION:
This study is an open Label, non-randomized, single-arm and multi-centered phase II clinical trial. It plans to evaluate the safety and efficacy of fruquintinib in advanced pancreatic cancer patients who failed second-line gemcitabine or 5-FU based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old;
2. Locally advanced or recurrent/metastatic pancreatic adenocarcinoma confirmed by cytological or histopathological examination;
3. Have failed second-line chemotherapy (gemcitabine or 5-FU-based regiments) (the definition of treatment failure is: toxic and side effects are intolerable, disease progression during treatment, recurrence within six months after the end of adjuvant chemotherapy, or progression within three months after the end of palliative chemotherapy); prior chemotherapy are required to include gemcitabine or 5-FU or its derivatives;
4. With one or more measurable lesions, the longest diameter should be at least 10 mm measured by spiral CT scan, or at least 20 mm by conventional CT scan should be(RECIST standard, version 1.1);
5. ECOG score was 0-2;
6. Life expectancy ≥12 weeks;
7. The damage was recovered from other antitumor treatments, including the interval from nitroso or mitomycin to enrollment was ≥6 weeks, and the interval from other cytotoxic drugs, radiotherapy or surgery to enrollment was ≥4 weeks, and the wound was completely healed;
8. Acceptable hematologic, hepatic, and renal function within 7 days from screenin: absolute neutrophil count (ANC) ≥1.5x109 /L; Hemoglobin ≥ 9.0g/dL; Platelet count ≥80 x109 /L; Total bilirubin < 1.5 times upper limit of normal (ULN); ALT and AST< 2.5 x ULN (with liver metastasis <5x ULN); Serum creatinine ≤1 x ULN, endogenous creatinine clearance rate >50ml/min;
9. Women of reproductive age need to take effective contraceptive measures;
10. Participate in this study is voluntarily and sign informed consent. With good compliance to cooperate with the follow-up, participate should understand the purpose of this study and the necessary procedures.

Exclusion Criteria:

1. A history of other malignant tumors in the past 5 year: however, localized tumor cured in the study is excluded, including cervical carcinoma in situ and skin basal cell carcinoma.
2. Patients with hypertension that could not be controlled by antihypertensive drug therapy (systolic blood pressure >140mmHg, diastolic blood pressure >90mmHg), coronary heart disease of grade 1 or above, arrhythmia of grade 1 or above (including prolonged QTc interval > 450ms in males and > 470ms in females) and cardiac dysfunction of grade 1 or above;
3. Symptomatic brain or meningeal metastases (except those with stable brain metastases for more than one month after treatment);
4. Have a history of uncontrolled epileptic seizures, central nervous system dysfunction, or mental disorders;
5. Uncontrolled pleural or abdominal effusion;
6. Undergoing kidney dialysis;
7. Severe or uncontrolled infection;
8. With multiple factors affecting oral medication (inability to swallow, chronic diarrhea and intestinal obstruction);
9. Abnormal coagulation function (PT>16s, APTT>43s, TT>21s, Fbg< 2g/L), bleeding tendency, receiving thrombolytic or anticoagulant treatment, and a history of thrombosis or embolism within six months;
10. Patients at risk of gastrointestinal bleeding should not be enrolled, including: (1) patients with active digestive ulcer lesions and fecal occult blood (2+ or above); (2) patients with history of black stools and hematemesis within 3 months; (3) Patients with gastrointestinal fistula or perforation.
11. Participated in other medicine clinical trials within four weeks.
12. Weight less than 40kg.
13. Urine protein ≥2+ by urine routine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
progression free survival (PFS) | up to 24 months
  The time from confirmation of enrollment to tumor progression or death from any cause, whichever came first

SECONDARY OUTCOMES:
overall survival (OS) | up to 36 months
  The time from randomization to death from any cause, whichever came first
objective response rate (ORR) | through study completion, an average of 2 year
  The proportion of patients whose tumors shrink to a certain extent and remain constant for a certain period of time
disease control rate (DCR) | through study completion, an average of 2 year
  percentage of cases with response to treatment (PR+CR) and disease stability (SD) that can be evaluated
duration of response (DoR) | through study completion, an average of 2 year
  the length of time that a tumor continues to respond to treatment without the cancer growing or spreading
safety: the potential side effects | through study completion, an average of 2 year
  the potential side effects

CONTACTS AND LOCATIONS:
Overall Officials: Weijian Guo, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li J, Qin S, Xu RH, Shen L, Xu J, Bai Y, Yang L, Deng Y, Chen ZD, Zhong H, Pan H, Guo W, Shu Y, Yuan Y, Zhou J, Xu N, Liu T, Ma D, Wu C, Cheng Y, Chen D, Li W, Sun S, Yu Z, Cao P, Chen H, Wang J, Wang S, Wang H, Fan S, Hua Y, Su W. Effect of Fruquintinib vs Placebo on Overall Survival in Patients With Previously Treated Metastatic Colorectal Cancer: The FRESCO Randomized Clinical Trial. JAMA. 2018 Jun 26;319(24):2486-2496. doi: 10.1001/jama.2018.7855. PMID 29946728
- [Result] Martin LK, Li X, Kleiber B, Ellison EC, Bloomston M, Zalupski M, Bekaii-Saab TS. VEGF remains an interesting target in advanced pancreas cancer (APCA): results of a multi-institutional phase II study of bevacizumab, gemcitabine, and infusional 5-fluorouracil in patients with APCA. Ann Oncol. 2012 Nov;23(11):2812-2820. doi: 10.1093/annonc/mds134. Epub 2012 Jul 5. PMID 22767582
- [Result] Rougier P, Riess H, Manges R, Karasek P, Humblet Y, Barone C, Santoro A, Assadourian S, Hatteville L, Philip PA. Randomised, placebo-controlled, double-blind, parallel-group phase III study evaluating aflibercept in patients receiving first-line treatment with gemcitabine for metastatic pancreatic cancer. Eur J Cancer. 2013 Aug;49(12):2633-42. doi: 10.1016/j.ejca.2013.04.002. Epub 2013 Apr 30. PMID 23642329
- [Result] Cao J, Zhang J, Peng W, Chen Z, Fan S, Su W, Li K, Li J. A Phase I study of safety and pharmacokinetics of fruquintinib, a novel selective inhibitor of vascular endothelial growth factor receptor-1, -2, and -3 tyrosine kinases in Chinese patients with advanced solid tumors. Cancer Chemother Pharmacol. 2016 Aug;78(2):259-69. doi: 10.1007/s00280-016-3069-8. Epub 2016 Jun 14. PMID 27299749